CLINICAL TRIAL: NCT00679393
Title: A Prospective Randomized Multicentre Clinical Trial Comparing Open Reduction Internal Fixation With Primary Subtalar Fusion in Patients With Severely Comminuted (Sanders IV), Displaced, Intra-articular Fractures of the Calcaneus
Brief Title: Comparative Study of Fixation or Fusion of Calcaneal Fractures
Acronym: Sanders IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Orthopaedic Trauma Association (Other); AO North America (Other)
Responsible Party: Principal Investigator, Richard Buckley, Clinical Professor, Section of Orthopaedics, Department of Surgery, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17526
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Fractures, Comminuted; Fracture Fixation, Internal
Keywords: Calcaneus; Intra-articular fracture; open reduction internal fixation; primary subtalar fusion
MeSH Terms: conditions — Fractures, Comminuted; Intra-Articular Fractures | interventions — Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fix (Other): Open reduction internal fixation of severely comminuted calcaneal fracture (Sanders IV)
  Interventions: Procedure: Open reduction internal fixation
- Fuse (Other): Primary subtalar fusion of severely comminuted calcaneal fractures (Sanders IV).
  Interventions: Procedure: Fusion

INTERVENTIONS:
Procedure: Open reduction internal fixation — Open reduction internal fixation surgery of severely comminuted calcaneal fracture (Sanders IV).
  Arms: Fix
Procedure: Fusion — Primary subtalar fusion of severely comminuted calcaneal fracture (Sanders IV)
  Arms: Fuse

SUMMARY:
A multicentre randomized controlled trial that will be conducted at Level 1 trauma centres across Canada. It will compare patients who receive open reduction, internal fixation for Sanders IV calcaneal fractures to patients who receive primary subtalar fusion for the same type of fracture. Patients will be followed up for a period of two years from the time of operation with evaluations being performed at 5 time points: 6 weeks, 3 months, 6 months, 12 months, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with Sanders IV displaced intra-articular calcaneal fracture
* males and females aged 16-59 inclusive
* ability to provide informed consent
* available for follow-up for at least 2 years after injury

Exclusion Criteria:

* medical contraindications to surgery
* previous calcaneal pathology (infection, tumor, etc)
* co-existent foot or ipsilateral lower limb injury
* open calcaneal fracture
* injury greater than 3 weeks old
* head injured patients
* inability to obtain pre-operative CT scan or accurately classify the fractures according to the Sanders classification system
* inability to comply with advice to diminish smoking after the injury
* metal allergy
* extremely comminuted intra-articular fractures of the calcaneus deemed impossible to reconstruct by the treating surgeon
* any concerns either by the treating surgeon or patient about harvesting autograft needed for fusion

Ages: 16 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2004-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
General Health Survey - SF-36 | 6 months, 12 months, and 24 months

SECONDARY OUTCOMES:
Validated Visual Analogue Scale | 6 months, 12 months, and 24 months
Musculoskeletal Function Assessment | 6 months, 12 months, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Buckley, MD, Principal Investigator — University of Calgary
Locations (4):
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - Halifax Infirmary, QEII Health Sciences Center, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario